CLINICAL TRIAL: NCT02673697
Title: Perceval Sutureless Implant Versus Standard-Aortic Valve Replacement A Controlled Randomized Trial in the Surgical Treatment of Aortic Valve Disease
Brief Title: Perceval Sutureless Implant Versus Standard-Aortic Valve Replacement
Acronym: PERSIST-AVR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Corcym S.r.l (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPS003
Record Dates: First submitted 2016-01-21; First posted 2016-02-04 (Estimated); Results first posted 2022-07-27 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Aortic Valve Disease; Aortic Stenosis
Keywords: Sutureless valve
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Perceval (Experimental): The Perceval sutureless aortic heart valve (Perceval valve) is a bioprosthesis manufactured with bovine pericardium and assembled on a Nitinol stent. The Perceval valve is designed to offer an alternative to surgically implanted flexible prostheses (stented and stentless biological valves). A special feature of the device is that it is self-anchoring and does not require sutures to be fixed to the implant site.
  Interventions: Device: Perceval valve
- other Stented biological valves (Active Comparator): The comparator will be other commercially approved standard biological sutured stented valves, both bovine and porcine. The choice of the comparator tissue valve will be at the discretion of the participating investigators.
  Interventions: Device: other stented biological valve

INTERVENTIONS:
Device: Perceval valve — Sutureless Aortic Biological Valve
  Arms: Perceval
Device: other stented biological valve — Any biological stented valves available on the market (Edwards, Medtronic, St.Jude, LivaNova, Labcor)
  Arms: other Stented biological valves

SUMMARY:
Prospective, randomized, stratified non blinded multi-center, international, post market trial assessed in a non-inferiority study.

The trial has a flexible sample size that will be determined adaptively. The trial will enroll up to 1234 subjects, but accrual may stop earlier at approximately 900 or 1050 subjects These subjects will be enrolled at approximately 60 worldwide investigational sites where the device is commercially available The primary objective of this trial is to test the safety and efficacy of Perceval versus standard sutured stented bioprosthetic aortic valves among the intended trial population.

DETAILED DESCRIPTION:
PERSIST-AVR is designed to collect data on sutureless valve (Perceval sutureless aortic heart valve), a new type of biological aortic valve, comparing data with standard biological aortic valve, considered the gold standard for aortic valve replacement. This prospective, randomized international multicenter study is planned to demonstrate, as primary endpoint, the non inferiority of Major Adverse Cardiac and Cerebrovascular (MACCE) events at one year while showing superiority in resource consumptions at hospital discharge in patients treated with Perceval valve when compared to standard aortic valve replacement. The study is planned to cover the lack of prospective, randomized comparison data between sutureless valve and standard aortic biological sutured valve. The trial has a flexible sample size that will be determined adaptively. The trial will enroll up to 1234 subjects, but accrual may stop earlier at approximately 900 or 1050 subjects. These subjects will be enrolled at approximately 60 worldwide investigational sites where the device is commercially available. The primary endpoint will be reached at 1 year FU and, consequently, the planned primary analysis will be performed 12 months following the end of accrual.

The be part of the trial, investigational sites should have demonstrated experience with the implantation of the Perceval and able to implement the requirements of the study protocol.. All subjects with severe symptomatic aortic stenosis or steno-insufficiency who are candidates for surgical replacement of their native aortic valve according to established guidelines in current medical practice and as specified in the Perceval valve Instruction for Use (IFU) are the intended population for inclusion in this randomized trial.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has an indication for treatment by valve replacement with a bioprosthesis according to the IFU, through either full sternotomy or mini-sternotomy.
2. The subject has aortic valve disease that can be treated with a commercially available Perceval valve size, based on preoperative CT-scan.
3. The subject has:

   1. critical aortic valve area defined as an initial aortic valve area of ≤1.0 cm2 or aortic valve area index < 0.6 cm2/m2 AND
   2. Mean gradient > 40 mmHg or Vmax > 4 m/sec by resting echocardiogram or simultaneous pressure recordings at cardiac catheterization [or with dobutamine stress, if subject has a left ventricular ejection fraction (LVEF) <55%] or velocity ratio < 0.25;
4. The subject is symptomatic due to aortic stenosis with functional class of New York Heart Association (NYHA) II or higher.
5. The subject has signed the informed consent.
6. The subject is of legal minimum age.
7. The subject will be available for postoperative follow-up beyond one year.

Exclusion Criteria:

1. The subject has a contraindication for treatment by the Perceval valve or by a bioprosthetic aortic valve as stated in the IFU.
2. The subject has aneurismal dilation or dissection of the ascending aortic wall.
3. The subject is scheduled for concomitant procedures other than Coronary Aortic Bypass Graft (CABG), myectomy with or without aortic annulus enlargement
4. The subject has congenital bicuspid (i.e. Sievers type 0) or unicuspid aortic valve.
5. Anatomical structures not suitable for Perceval valve such as: aortic root enlargement, where the ratio between the diameter of the sino-tubular junction and the annulus diameter is > 1.3.
6. The subject has a prosthetic heart valve in any position, including mitral valve repair.
7. The subject has a stroke or myocardial infarction (STEMI and NSTEMI) within 30 days prior to the planned valve implant surgery.
8. The subject has active endocarditis, myocarditis, or sepsis.
9. The subject is in cardiogenic shock manifested by low cardiac output and needing hemodynamic support.
10. The subject is allergic to nickel alloys.
11. The subject is already included in another clinical trial that could confound the results of this clinical investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 914 (Actual)
Dates: Start 2016-03-22 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodor Fischlein, MD, Principal Investigator — Klinikum Nurnberg, Nurnberg, Germany; Roberto Lorusso, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (47):
- United States (5):
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - Maine Medical Center, Portland, Maine
  - Heart and Vascular Institute, Cleveland Clinic, Cleveland, Ohio
  - Houston Methodist Research Institute, Houston Methodist Hospital, Houston, Texas
  - Valley Health System, Winchester, Virginia
- Austria (4):
  - Klinische Abteilung fuer Herzchirurgie, Graz
  - Medical University of Innsbruck, Innsbruck
  - Herzzentrum Hietzing, Vienna
  - Medical University of Vienna, Vienna
- Belgium (3):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Cliniques Univ. Saint-Luc, Brussels
  - Universitair Ziekenhuis, Leuven
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec
- Hospital Clinico San Borja Arriaran, Santiago, Chile
- France (7):
  - CHU Angers, Angers
  - C.H.U. de Besançon, Besançon
  - Hôpital privé de Bois Bernard, Bois-Bernard
  - Chru De Lille, Lille
  - CHU Arnaud de Villeneuve, Montpellier
  - C.H.U. de Nancy, Nancy
  - CHU de Poitiers, Poitiers
- Germany (7):
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Herz- und Gefäß-Klinik, Bad Neustadt an der Saale
  - Herzzentrum Dresden GmbH Universitätsklinik, Dresden
  - ASKLEPIOS Klinikum Harburg, Hamburg
  - University Heart Center Hamburg, Hamburg
  - Medizinische Hochschule, Hanover
  - Klinikum Nürnberg, Nuremberg
- Israel (2):
  - Shaare Zedek Medical Center, Jerusalem
  - Sheba medical Center, Tel Aviv
- Italy (8):
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia, BS
  - Centro Cuore Morgagni Pedara, Pedara, CT
  - Ospedale San Raffaele, Milan, MI
  - lstituto Clinico Sant'Ambrogio e San Siro, Milan, MI
  - Fondazione Toscana Gabriele Monasterio-Presidio Ospedaliero di Massa, Massa, MS
  - Spedali Civili, Brescia
  - Maria Cecilia Hospital, Cotignola
  - Azienda Ospedaliera Carlo Poma, Mantova
- Netherlands (2):
  - Catharina Ziekenhuis, Eindhoven
  - Maastricht University Hospital, Maastricht
- Spain (3):
  - Complejo Hospitalario Universitario De A Coruña, A Coruña
  - Hospital University Germans Trias I Pujol, Badalona
  - Hospital Clinico Universitario Virgen De La Arrixaca, Murcia
- Victoria Hospital, Blackpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lorusso R, Folliguet T, Shrestha M, Meuris B, Kappetein AP, Roselli E, Klersy C, Nozza M, Verhees L, Larracas C, Goisis G, Fischlein T. Sutureless versus Stented Bioprostheses for Aortic Valve Replacement: The Randomized PERSIST-AVR Study Design. Thorac Cardiovasc Surg. 2020 Mar;68(2):114-123. doi: 10.1055/s-0038-1675847. Epub 2018 Nov 29. PMID 30497085
- [Result] Fischlein T, Folliguet T, Meuris B, Shrestha ML, Roselli EE, McGlothlin A, Kappert U, Pfeiffer S, Corbi P, Lorusso R; Perceval Sutureless Implant Versus Standard-Aortic Valve Replacement Investigators. Sutureless versus conventional bioprostheses for aortic valve replacement in severe symptomatic aortic valve stenosis. J Thorac Cardiovasc Surg. 2021 Mar;161(3):920-932. doi: 10.1016/j.jtcvs.2020.11.162. Epub 2020 Dec 14. PMID 33478837
- [Derived] Lorusso R, Ravaux JM, Pollari F, Folliguet TA, Kappert U, Meuris B, Shrestha ML, Roselli EE, Bonaros N, Fabre O, Corbi P, Troise G, Andreas M, Pinaud F, Pfeiffer S, Kueri S, Tan E, Voisine P, Girdauskas E, Rega F, Garcia-Puente J, Fischlein T; on behalf the PERSIST-AVR Investigators. Pacemaker implantation after sutureless or stented valve: results from a controlled randomized trial. Eur J Cardiothorac Surg. 2022 Sep 2;62(4):ezac164. doi: 10.1093/ejcts/ezac164. PMID 35290444
- [Derived] Lorusso R, Jiritano F, Roselli E, Shrestha M, Folliguet T, Meuris B, Pollari F, Fischlein T; PERSIST-AVR Investigators. Perioperative platelet reduction after sutureless or stented valve implantation: results from the PERSIST-AVR controlled randomized trial. Eur J Cardiothorac Surg. 2021 Dec 1;60(6):1359-1365. doi: 10.1093/ejcts/ezab175. PMID 34118150

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 914 patients were enrolled in the PERSIST-AVR trial. Among the 914 patients enrolled, 910 underwent randomization
Pre-assignment Details: A total of 914 patients were enrolled in the PERSIST-AVR trial. Among the 914 patients enrolled, 910 underwent randomization. 4 patients were not randomized due to consent withdrawal (2 cases) and physician decision (2 cases)
Period: Overall Study
Arm/Group | Perceval | Other Stented Biological Valves
Started (Randomized) | 453 | 457
Implanted | 450 | 446
Per-Protocol Population | 407 | 412
Completed | 0 | 0
Not Completed | 453 | 457
Not completed — Adverse Event | 2 | 0
Not completed — Death | 32 | 24
Not completed — Lost to Follow-up | 5 | 2
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 10 | 7
Not completed — Change subj medical status | 1 | 2
Not completed — Explant | 10 | 5
Not completed — Sponsor Decision to stop follow up | 391 | 416

BASELINE CHARACTERISTICS:
Population: Per Protocol Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Perceval | Other Stented Biological Valves | Total
Number analyzed (Participants) | 407 | 412 | 819
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.4 (5.6) | 75.0 (6.1) | 75.2 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204 | 185 | 389
  Male | 203 | 227 | 430
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Freedom From Major Adverse Cardiac and Cerebrovascular Events (MACCE)
Description: The primary endpoint is freedom from MACCE (composite endpoint of all cause death, myocardial infarction, stroke, and valve re-intervention) at one year based on Clinical Event Committee (CEC) adjudication.
Time Frame: 1 year post-operatively
Population: Per Protocol Population
Measure: Mean (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Perceval | Other Stented Biological Valves
Number analyzed (Participants) | 407 | 412
Proportion of participants | 0.917 [0.888 to 0.942] | 0.920 [0.892 to 0.945]
Statistical Analysis 1: Comparison: Perceval vs Other Stented Biological Valves; A the primary analysis will compare Perceval valve (Treatment arm) vs. standard sutured stented valve (Control arm) on the Per Protocol population. A one-sided non-inferiority test, using the non-inferiority margin Δ=0.05, will be performed to compare the two arms on the proportion of subjects that are event-free at one year (primary analysis); Test type: Non-Inferiority — The primary analysis will calculate the Bayesian posterior probability that the difference [MACCECONTROL - MACCEPERCEVAL] is lower than 0.05 (predetermined non-inferiority margin): The null hypothesis will be rejected, and non-inferiority concluded, if the posterior probability exceeds 0.9775 at the final analysis; p = 0.9914, Bayesian — The null hypothesis will be rejected, and non-inferiority concluded, if the posterior probability exceeds 0.9775 at the final analysis

2. Secondary Outcome: Surgical Times
Description: 1. Cross clamp time during index procedure
  2. Cardiopulmonary bypass time during index procedure
  Start time and finish time were collected for operative room time procedure and calculated for each subject. Mean was calculated and reported in the results sections
Time Frame: Intra-operative
Population: Safety population (actual treatment)
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Perceval | Other Stented Biological Valves
Number analyzed (Participants) | 450 | 446
Minutes
  Cardiopulmonary bypass time | 71.0 (34.1) | 87.8 (33.9)
  Cross clamp time | 48.5 (24.7) | 65.2 (23.6)

ADVERSE EVENTS:
Time Frame: All serious adverse events were collected from implant to study closure (2 years completed) (July 31, 2020)
Description: The Principal investigator was required to report to the Sponsor:
  * all serious adverse events (SAE)
  * all device deficiencies
  * all Unanticipated Serious Adverse Device Effects (USADE)
  Incidences of events are here reported for the Safety Population (actual treatment) based on Clinical Event Commitee Adjudication
Arm/Group | Perceval | Other Stented Biological Valves
All-Cause Mortality (participants affected / at risk) | 32/450 | 24/446
Serious Adverse Events (participants affected / at risk) | 390/450 | 342/446
Other Adverse Events (participants affected / at risk) | 0/450 | 0/446
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perceval (N=450) | Other Stented Biological Valves (N=446)
Myocardial Infarction (Cardiac disorders) | 6 (7) | 15 (16)
Stroke (Nervous system disorders) | 21 (22) | 16 (16)
Aortic valve re-intervention (Cardiac disorders) | 13 (13) | 7 (7)
Transient Ischemic Attack (Nervous system disorders) | 7 (8) | 4 (4)
Bleeding (Vascular disorders) | 30 (31) | 39 (44)
Acute Kidney Injury (Renal and urinary disorders) | 10 (10) | 13 (15)
Endocarditis (Cardiac disorders) | 11 (14) | 15 (17)
Structural Valve Deterioration (Cardiac disorders) | 2 (3) | 1 (1)
Valve thrombosis (Cardiac disorders) | 2 (2) | 0 (0)
Arrhythmia or conduction disorder (Cardiac disorders) | 100 (102) | 76 (87)
Thromboembolic event, non-cerebral (Vascular disorders) | 3 (3) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (11) | 2 (2)
Major vascular complication (Vascular disorders) | 3 (3) | 3 (3)
Other cardiovascular SAE (Vascular disorders) | 39 (43) | 26 (28)
Other non-cardiovascular SAE (General disorders) | 132 (171) | 121 (170)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/97/NCT02673697/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT02673697/SAP_001.pdf